CLINICAL TRIAL: NCT03322670
Title: Description of Pneumococcal Community-acquired Pneumonia in General Practice in France
Brief Title: Description of Pneumococcal Pneumonia
Acronym: PneumoCAP
Status: Completed | Type: Observational
Sponsor: CNGE Conseil (Other)
Responsible Party: Principal Investigator, GILBERG SERGE, Professor of Family practice, CNGE Conseil
Other Study IDs: N° ID RCB : 2016-A01537-44
Record Dates: First submitted 2017-09-25; First posted 2017-10-26 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Community-acquired Pneumonia
Keywords: community-acquired pneumonia; family practice; streptococcus pneumoniae
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood:
    * Blood count
    * CRP
    * Procalcitonin (PCT)
    * Blood cultures
  * Oropharynx:
    - Oropharyngeal sample: for multiplex polymerase chain reaction (PCR)
  * Sputum:
    - Sputum sample testing (induced expectoration if possible)
  * Urine:
    * Pneumococcal urinary antigen test (Alere BinaxNOW)
    * Luminex technology-based multiplex urine antigen detection (UAD)
    * Urine collection (for urine bank at Central Laboratory)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Signs of CAP and a positive chest X-Ray: Patients with at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization) and and a chest X-Ray not compatible with CAP
  Interventions: Other: Signs of CAP and a positive chest X-Ray
- Patients directly hospitalized: Patients with at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization) and and who are directly hospitalized before complementary examinations
  Interventions: Other: Patients directly hospitalized
- Control patients: Healthy Patients (age-matched with a radiologically confirmed CAP patient)
  Interventions: Diagnostic Test: Control patients
- Patients with partial participation: Patients with at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization) and who can not or do not want to perform all the complementary examinations of the study
  Interventions: Other: Patients with partial participation
- Signs of CAP and a negative Chest X-Ray: Patients with at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization) and and a chest X-Ray not compatible with CAP
  Interventions: Other: Signs of CAP and a negative chest X-Ray

INTERVENTIONS:
Other: Signs of CAP and a positive chest X-Ray — * collection of clinical examination data
  * biological and bacteriological examinations (blood, urine, sputum, nasopharyngeal)
  * self-reported questionnaires on duration of symptoms and restriction of activity
  * telephone contact on day 28 and day 90 if hospitalized before day 28
  Groups: Signs of CAP and a positive chest X-Ray
Other: Patients directly hospitalized — * collection of clinical examination data
  * telephone contact on day 28 and retrieval of hospitalization report
  * telephone contact on day 90
  Groups: Patients directly hospitalized
Diagnostic Test: Control patients — - bacteriological examinations (urine)
  Groups: Control patients
Other: Patients with partial participation — - collection of clinical examination data
  Groups: Patients with partial participation
Other: Signs of CAP and a negative chest X-Ray — * collection of clinical examination data
  * telephone contact on day 28
  Groups: Signs of CAP and a negative Chest X-Ray

SUMMARY:
Statement of the problem:

Overprescription of antibiotics raises important public health issues because of the emergence of multiresistant bacteria by selection pressure. The results of the observational prospective study entitled "CAPA" on the description of 886 suspected cases of acute community-acquired pneumonia (CAP) treated in general practices in France confirm that, whatever the etiologic hypothesis and the results of the chest X-ray, these patients routinely receive antibiotics. Therefore, it is important to be able to distinguish cases of pneumococcal CAP in which early antibiotic treatment is justified from those cases for which another strategy could be considered.

Primary objective:

To identify the clinical, biological and radiological characteristics of patients with pneumococcal CAP amongst all patients with CAP radiologically confirmed, in general practice in France.

Design :

Prospective cross-sectional descriptive study.

Inclusion criteria. Adults older than 18 showing clinical signs suggestive of CAP (at least one sign of infection and at least one pulmonary sign) and able to realize chest X ray within 6 hours after prescription.

Patient follow-up procedures. Patients will be treated by standard of care according to French recommendations. After observing clinical signs suggestive of CAP, the physician prescribes a chest X-ray. Then, protocol-specific examinations (blood sample, oropharyngeal sample for multiplex polymerase chain reaction (PCR), sputum sample testing (induced expectoration if possible), urinary sample) will be performed on all out patients. Patients will be contacted again on day 28 to increase diagnostic certainty. For patients with clinical signs of CAP and hospitalized, the investigator will ask their consent to retrieve the hospital report, on or before day 28 and to be contacted on day 90.

DETAILED DESCRIPTION:
The aim of the study is to enroll approximately 2000 patients with CAP in total. Approximately 1000 X-ray positive patients and 1000 X-ray negative patients will be enrolled over 18 months.

Investigating GPs will identify patients with clinical signs suggestive of CAP at clinic visits.

A chest X-ray will be prescribed in accordance with local standard of care practices for patients that do not require immediate hospitalization. Chest X-ray must be completed within the 6 hours following its prescription.

For the 1000 patients (patient enrolment will be monitored centrally) with a positive chest X-ray, all procedures will be undertaken according to the protocol. Patients will attend the local medical analysis laboratory for biological sample collection (blood, sputum, oropharyngeal swab for the PCR, and urine). If a patient has taken antibiotics prior to the clinic visit at which CAP is suspected, will only have urine samples collected.

As a diagnostic confirmation of the chest X-ray assessments, for the 1000 patients for whom the local radiologist will have diagnosed a parenchymal opacity compatible with CAP, 200 patients will be randomly selected by the clinical research organization (CRO Paris Descartes Necker Cochin). A central independent thoracic radiologist expert will re-read their chest X-ray. In case of insufficient agreement, all chest X-rays will be re-read.

Patients will be asked to complete and return a self-assessment questionnaire at day 7 (D7) and at day 14 (D14) on the number of work days missed, if any, interruption of occupational activity, and the number of days of restricted everyday activities or recreational.

Patients will be contacted by telephone at day 28, and day 90 if they are hospitalized between day 0 and day 28.

For the 1000 patients (patient enrolment will be monitored centrally) with a negative chest X-ray, no medical analysis will be performed. Only clinical examination data will be recorded. Patients will be contacted by telephone at day 28.

For patients who will be directly hospitalized before the completion of the additional examinations, they will be contacted by telephone at day 28 to retrieve the hospitalization report and at day 90.

Control Patients will be included for the assessment of Pneumococcal urine antigen detection (UAD) Assay: in the two weeks following the inclusion of a patient with CAP, investigators should include a control patient according to the control patient inclusion / exclusion criteria. For these healthy patients, the number of inclusion is limited to 400.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria for suspected CAP population:

* Age ≥18 years
* Presence of at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization):

  * at least one sign of infection

    * fever > 38.5°C (maximum temperature measured by the patient or GP)
    * tachycardia > 100 /min
    * hyperpnea > 20/min
    * global impression of severity*
    * muscle aches, fatigue, or chills
  * and at least one sign of pulmonary localization

    * cough
    * unilateral chest pain
    * purulent or non-purulent sputum
    * auscultatory abnormality compatible with CAP (focus of crackles)
* Affiliation with health insurance system
* Chest X-ray performed within 6 hours of presenting to the general practice
* Willing and capable of providing blood, oropharyngeal urine samples, and sputum sample, for filling self-administered questionnaires to D7 and D14 and to be contacted again on D28 and on D90 if necessary, if chest X-ray is positive.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.

  * Inclusion criteria for who do not wish to participate in the full study or who have not received a chest X-ray
* Age ≥18 years
* Presence of at least 2 signs suggestive of CAP on presentation at general practice (one general sign of infection and one sign of pulmonary localization):

  * at least one sign of infection

    * fever > 38.5°C (maximum temperature measured by the patient or GP)
    * tachycardia > 100 /min
    * hyperpnea > 20/min
    * global impression of severity*
    * muscle aches, fatigue, or chills
  * and at least one sign of pulmonary localization

    * cough
    * unilateral chest pain
    * purulent or non-purulent sputum
    * auscultatory abnormality compatible with CAP (focus of crackles)
    * Control Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* A signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Age ≥18 years.
* Patients who are will to provide a urine sample

Exclusion Criteria:

* Exclusion criteria for suspected CAP population:

  * conditions of medical treatment not allowing for chest X-ray within 6 hours after diagnosis of CAP
  * contraindication to chest X-ray
  * conditions of medical management not allowing the realization of biological and bacteriological examinations within 8 hours of D0 consultation (except for patient immediately hospitalized)
  * chest X-ray finding not compatible with CAP : chest X-ray showing another lung disease than a CAP (for example: pulmonary neoplasia, tuberculosis, pulmonary embolism)
* Control Exclusion Criteria

Patients presenting with any of the following will not be included in the study:

* Patients who are investigational site staff members or relatives of those site staff member or subjects who are Pfizer employees directly involved in the conduct of the trial.
* Patients with suspicion of CAP or other respiratory infectious diseases, as well as evidence of or documented concomitant infectious disease.
* Patients residing in any long-term care facilities (for example, nursing homes, respite care facilities, etc).
* Patients with known bronchial obstruction or a history of post-obstructive pneumonia. Chronic obstructive pulmonary disease (COPD) is permissible, provided there has not been an exacerbation within the 3 months prior to enrollment.
* Patients with primary lung cancer or another malignancy metastatic to the lungs.
* Patients with fever (measured temperature of ≥38.0° C measured by a healthcare provider).
* Patients with significant immunosuppressive disease such as AIDS, leukemia, etc.
* Patients with either pneumococcal conjugate vaccine (PCV) and/or pneumococcal polysaccharide vaccine (PPV) administration within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In France, patients who visit a General Practitioner and who have clinical signs suggestive of CAP at clinic visits.
  For the control cohort, healthy patient who visit a General Practitioner in the two weeks following the inclusion of a patient with CAP confirmed on the chest X-ray
Sampling Method: Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Percentage of pneumococcal CAP amongst the other etiological CAP with a positive chest X-ray | Day 0
  Determination oh the proportion of pneumococcal CAP among all CAP radiologically confirmed with other etiologies identified, followed in general practice in France. Comparison of the clinical, biological and radiological characteristics of patients with radiologically confirmed pneumococcal CAP to those with radiologically confirmed CAP patients for whom another microbiological etiology was identified

SECONDARY OUTCOMES:
Description of clinical characteristics of patients treated in general practice for a radiologically confirmed CAP, based on the microbiological etiologies | Day 0
  Number and percentage of each of the clinical characteristics according to the microbiological etiology according to the presence or not of a sepsis and according to an hospitalization or not

OTHER OUTCOMES:
Description of biological characteristics of patients treated in general practice for a radiologically confirmed CAP, based on the microbiological etiologies | Day 0
  Number and percentage of each of the biological characteristics according to the microbiological etiology according to the presence or not of a sepsis and according to an hospitalization or not
Description radiological characteristics of patients treated in general practice for a radiologically confirmed CAP, based on all the microbiological etiologies. | day 0
  Number and percentage of each of the radiological characteristics according to the microbiological etiology according to the presence or not of a sepsis and according to an hospitalization or not
Incidence rate of pneumococcal CAP radiologically confirmed on chest X-ray, in the general practitioners settings | Day 0
  Number of adult patients with pneumococcal CAP and positive chest X-Ray and the number of adult patients with clinical signs of CAP (defined as 2 signs suggestive of CAP) in general practice
Descriptive analysis of Streptococcus pneumoniae serotypes identified on the urine assays. | Day 0
  Number of pneumonia according to each serotype of Streptococcus pneumoniae identified on the Urine Antigen Detection, among all pneumococcal CAP
Descriptive analysis of Streptococcus pneumoniae serotypes identified on the blood culture | Day 0
  Number of pneumonia according to each serotype of Streptococcus pneumoniae identified on the blood culture, among all pneumococcal CAP
Descriptive analysis of Streptococcus pneumoniae serotypes identified on the sputum culture | Day 0
  Number of pneumonia according to each serotype of Streptococcus pneumoniae identified on the sputum culture, among all pneumococcal CAP
Assessment of costs generated by pneumococcal CAP managed in ambulatory setting. | Day 90
  Costs of medical care (medical consultation, medicated treatment, hospitalization costs, work stoppage)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gilberg, Professor, Principal Investigator — University Paris Descartes
Locations (1):
- URC-CIC Paris Descartes-Cochin-Necker, Paris, France

REFERENCES:
- [Background] Hosker H, Cooke NJ, Hawkey P. Antibiotics in chronic obstructive pulmonary disease. BMJ. 1994 Apr 2;308(6933):871-2. doi: 10.1136/bmj.308.6933.871. No abstract available. PMID 8173363
- [Background] Wipf JE, Lipsky BA, Hirschmann JV, Boyko EJ, Takasugi J, Peugeot RL, Davis CL. Diagnosing pneumonia by physical examination: relevant or relic? Arch Intern Med. 1999 May 24;159(10):1082-7. doi: 10.1001/archinte.159.10.1082. PMID 10335685
- [Background] Jackson ML, Neuzil KM, Thompson WW, Shay DK, Yu O, Hanson CA, Jackson LA. The burden of community-acquired pneumonia in seniors: results of a population-based study. Clin Infect Dis. 2004 Dec 1;39(11):1642-50. doi: 10.1086/425615. Epub 2004 Nov 8. PMID 15578365
- [Background] Holm A, Nexoe J, Bistrup LA, Pedersen SS, Obel N, Nielsen LP, Pedersen C. Aetiology and prediction of pneumonia in lower respiratory tract infection in primary care. Br J Gen Pract. 2007 Jul;57(540):547-54. PMID 17727747
- [Background] Porath A, Schlaeffer F, Lieberman D. The epidemiology of community-acquired pneumonia among hospitalized adults. J Infect. 1997 Jan;34(1):41-8. doi: 10.1016/s0163-4453(97)80008-4. PMID 9120323
- [Background] Said MA, Johnson HL, Nonyane BA, Deloria-Knoll M, O'Brien KL; AGEDD Adult Pneumococcal Burden Study Team; Andreo F, Beovic B, Blanco S, Boersma WG, Boulware DR, Butler JC, Carratala J, Chang FY, Charles PG, Diaz AA, Dominguez J, Ehara N, Endeman H, Falco V, Falguera M, Fukushima K, Garcia-Vidal C, Genne D, Guchev IA, Gutierrez F, Hernes SS, Hoepelman AI, Hohenthal U, Johansson N, Kolek V, Kozlov RS, Lauderdale TL, Marekovic I, Masia M, Matta MA, Miro O, Murdoch DR, Nuermberger E, Paolini R, Perello R, Snijders D, Plecko V, Sorde R, Stralin K, van der Eerden MM, Vila-Corcoles A, Watt JP. Estimating the burden of pneumococcal pneumonia among adults: a systematic review and meta-analysis of diagnostic techniques. PLoS One. 2013;8(4):e60273. doi: 10.1371/journal.pone.0060273. Epub 2013 Apr 2. PMID 23565216
- [Background] Musher DM, Thorner AR. Community-acquired pneumonia. N Engl J Med. 2014 Oct 23;371(17):1619-28. doi: 10.1056/NEJMra1312885. No abstract available. PMID 25337751
- [Background] Dorca J, Torres A. Lower respiratory tract infections in the community: towards a more rational approach. Eur Respir J. 1996 Aug;9(8):1588-9. doi: 10.1183/09031936.96.09081588. No abstract available. PMID 8866576
- [Background] Gennis P, Gallagher J, Falvo C, Baker S, Than W. Clinical criteria for the detection of pneumonia in adults: guidelines for ordering chest roentgenograms in the emergency department. J Emerg Med. 1989 May-Jun;7(3):263-8. doi: 10.1016/0736-4679(89)90358-2. PMID 2745948
- [Background] Metlay JP, Fine MJ. Testing strategies in the initial management of patients with community-acquired pneumonia. Ann Intern Med. 2003 Jan 21;138(2):109-18. doi: 10.7326/0003-4819-138-2-200301210-00012. PMID 12529093
- [Background] Partouche H, Buffel du Vaure C, Personne V, Le Cossec C, Garcin C, Lorenzo A, Ghasarossian C, Landais P, Toubiana L, Gilberg S. Suspected community-acquired pneumonia in an ambulatory setting (CAPA): a French prospective observational cohort study in general practice. NPJ Prim Care Respir Med. 2015 Mar 12;25:15010. doi: 10.1038/npjpcrm.2015.10. PMID 25763466
- [Background] Young M, Marrie TJ. Interobserver variability in the interpretation of chest roentgenograms of patients with possible pneumonia. Arch Intern Med. 1994 Dec 12-26;154(23):2729-32. doi: 10.1001/archinte.1994.00420230122014. PMID 7993157
- [Background] Claessens YE, Debray MP, Tubach F, Brun AL, Rammaert B, Hausfater P, Naccache JM, Ray P, Choquet C, Carette MF, Mayaud C, Leport C, Duval X. Early Chest Computed Tomography Scan to Assist Diagnosis and Guide Treatment Decision for Suspected Community-acquired Pneumonia. Am J Respir Crit Care Med. 2015 Oct 15;192(8):974-82. doi: 10.1164/rccm.201501-0017OC. PMID 26168322
- [Background] Ortqvist A, Hedlund J, Wretlind B, Carlstrom A, Kalin M. Diagnostic and prognostic value of interleukin-6 and C-reactive protein in community-acquired pneumonia. Scand J Infect Dis. 1995;27(5):457-62. doi: 10.3109/00365549509047046. PMID 8588135
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Le Bel J, Hausfater P, Chenevier-Gobeaux C, Blanc FX, Benjoar M, Ficko C, Ray P, Choquet C, Duval X, Claessens YE; ESCAPED study group. Diagnostic accuracy of C-reactive protein and procalcitonin in suspected community-acquired pneumonia adults visiting emergency department and having a systematic thoracic CT scan. Crit Care. 2015 Oct 16;19:366. doi: 10.1186/s13054-015-1083-6. PMID 26472401
- [Background] van Vugt SF, Broekhuizen BD, Lammens C, Zuithoff NP, de Jong PA, Coenen S, Ieven M, Butler CC, Goossens H, Little P, Verheij TJ; GRACE consortium. Use of serum C reactive protein and procalcitonin concentrations in addition to symptoms and signs to predict pneumonia in patients presenting to primary care with acute cough: diagnostic study. BMJ. 2013 Apr 30;346:f2450. doi: 10.1136/bmj.f2450. PMID 23633005
- [Background] van der Meer V, Neven AK, van den Broek PJ, Assendelft WJ. Diagnostic value of C reactive protein in infections of the lower respiratory tract: systematic review. BMJ. 2005 Jul 2;331(7507):26. doi: 10.1136/bmj.38483.478183.EB. Epub 2005 Jun 24. PMID 15979984
- [Background] Holm A, Pedersen SS, Nexoe J, Obel N, Nielsen LP, Koldkjaer O, Pedersen C. Procalcitonin versus C-reactive protein for predicting pneumonia in adults with lower respiratory tract infection in primary care. Br J Gen Pract. 2007 Jul;57(540):555-60. PMID 17727748
- [Background] Niederman MS. Biological markers to determine eligibility in trials for community-acquired pneumonia: a focus on procalcitonin. Clin Infect Dis. 2008 Dec 1;47 Suppl 3:S127-32. doi: 10.1086/591393. PMID 18986278
- [Background] Melbye H, Stocks N. Point of care testing for C-reactive protein - a new path for Australian GPs? Aust Fam Physician. 2006 Jul;35(7):513-7. PMID 16820825
- [Background] Christ-Crain M, Muller B. Procalcitonin and pneumonia: is it a useful marker? Curr Infect Dis Rep. 2007 May;9(3):233-40. doi: 10.1007/s11908-007-0037-9. PMID 17430706
- [Background] Roson B, Fernandez-Sabe N, Carratala J, Verdaguer R, Dorca J, Manresa F, Gudiol F. Contribution of a urinary antigen assay (Binax NOW) to the early diagnosis of pneumococcal pneumonia. Clin Infect Dis. 2004 Jan 15;38(2):222-6. doi: 10.1086/380639. Epub 2003 Dec 18. PMID 14699454
- [Background] Guchev IA, Yu VL, Sinopalnikov A, Klochkov OI, Kozlov RS, Stratchounski LS. Management of nonsevere pneumonia in military trainees with the urinary antigen test for Streptococcus pneumoniae: an innovative approach to targeted therapy. Clin Infect Dis. 2005 Jun 1;40(11):1608-16. doi: 10.1086/429919. Epub 2005 May 2. PMID 15889358
- [Background] Song JY, Eun BW, Nahm MH. Diagnosis of pneumococcal pneumonia: current pitfalls and the way forward. Infect Chemother. 2013 Dec;45(4):351-66. doi: 10.3947/ic.2013.45.4.351. Epub 2013 Dec 27. PMID 24475349
- [Background] Pride MW, Huijts SM, Wu K, Souza V, Passador S, Tinder C, Song E, Elfassy A, McNeil L, Menton R, French R, Callahan J, Webber C, Gruber WC, Bonten MJ, Jansen KU. Validation of an immunodiagnostic assay for detection of 13 Streptococcus pneumoniae serotype-specific polysaccharides in human urine. Clin Vaccine Immunol. 2012 Aug;19(8):1131-41. doi: 10.1128/CVI.00064-12. Epub 2012 Jun 6. PMID 22675155
- [Background] Reddington K, Tuite N, Barry T, O'Grady J, Zumla A. Advances in multiparametric molecular diagnostics technologies for respiratory tract infections. Curr Opin Pulm Med. 2013 May;19(3):298-304. doi: 10.1097/MCP.0b013e32835f1b32. PMID 23425918
- [Background] Jain S, Self WH, Wunderink RG, Fakhran S, Balk R, Bramley AM, Reed C, Grijalva CG, Anderson EJ, Courtney DM, Chappell JD, Qi C, Hart EM, Carroll F, Trabue C, Donnelly HK, Williams DJ, Zhu Y, Arnold SR, Ampofo K, Waterer GW, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, McCullers JA, Pavia AT, Edwards KM, Finelli L; CDC EPIC Study Team. Community-Acquired Pneumonia Requiring Hospitalization among U.S. Adults. N Engl J Med. 2015 Jul 30;373(5):415-27. doi: 10.1056/NEJMoa1500245. Epub 2015 Jul 14. PMID 26172429
- [Background] Houck PM, Bratzler DW, Nsa W, Ma A, Bartlett JG. Timing of antibiotic administration and outcomes for Medicare patients hospitalized with community-acquired pneumonia. Arch Intern Med. 2004 Mar 22;164(6):637-44. doi: 10.1001/archinte.164.6.637. PMID 15037492
- [Background] Flamaing J, De Backer W, Van Laethem Y, Heijmans S, Mignon A. Pneumococcal lower respiratory tract infections in adults: an observational case-control study in primary care in Belgium. BMC Fam Pract. 2015 May 27;16:66. doi: 10.1186/s12875-015-0282-1. PMID 26012956
- See also: Related Info — http://social-sante.gouv.fr/prevention-en-sante/preserver-sa-sante/calendrier-vaccinal